CLINICAL TRIAL: NCT02433158
Title: An Open-Label Extension Study to Evaluate the Safety of Rivipansel (GMI-1070) in the Treatment of One or More Vaso-Occlusive Crises in Hospitalized Subjects With Sickle Cell Disease
Brief Title: Safety of Rivipansel (GMI-1070) in the Treatment of One or More Vaso-Occlusive Crises in Hospitalized Subjects With Sickle Cell Disease
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The B5201003 OLE study was terminated based on the failure of the 'parent" B5201002 study to meet its efficacy endpoints. Termination was not due to safety.
Sponsor: GlycoMimetics Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B5201003
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Sickle Cell Anemia; Sickle Cell Disease; Sickle Cell Disorders; Pain Crisis; Vaso-occlusive Crisis
Keywords: Rivipansel; GMI-1070; Selectin Inhibitor; SCD; VOC
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — rivipansel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Includes one adult stratum (>18 years old) and one pediatric stratum (12-17 years old). Subjects aged 12 and over who weigh >40 kg, will receive a loading dose of 1680 mg followed by a maintenance dose of 840 mg.
  Interventions: Drug: Rivipansel
- Cohort 2 (Experimental): Includes one pediatric stratum (6-11 years old). Subjects 6 to 11 years of age or subjects who weigh 40 kg, will receive a loading dose of 40 mg/kg (maximum of 1680 mg) followed by a maintenance dose of 20 mg/kg (maximum of 840 mg).
  Interventions: Drug: Rivipansel

INTERVENTIONS:
Drug: Rivipansel — Rivipansel will be infused intravenously every 12 hours up to a maximum of 15 doses.
  Other Names: GMI-1070

SUMMARY:
This is an open label extension study in subjects with Sickle Cell Disease (SCD) who have completed the double blind Phase 3 study (B5201002).

DETAILED DESCRIPTION:
This is an open label extension study in subjects who are 6 years of age or older with Sickle Cell Disease (SCD) who have completed the double blind Phase 3 study (B5201002). This study is designed to evaluate the safety and describe the efficacy of rivipansel as treatment for one or more vaso-occlusive crisis (VOC) events in hospitalized subjects with SCD.

ELIGIBILITY:
Inclusion Criteria:

* Completion of Study B5201002.
* Documented diagnosis of SCD.
* At least 6 years of age.
* Male and female subjects of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study.
* Diagnosis of VOC necessitating IV opioids and admission to the hospital.
* Able to receive the first dose of rivipansel within 24 hours from administration of the first dose of IV opioids for this hospitalization.

Exclusion Criteria:

* Non-compliance with study procedures in the double blind study (B5201002).
* Occurrence of any severe and/or generalized cutaneous manifestation or any other adverse event during participation in Study B5201002 that was related to study drug and which would therefore make it inappropriate for the subject to receive rivipansel in the current study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results.
* Clinically significant deterioration in renal function in Study B5201002.
* Pregnant female subjects, breastfeeding female subjects and male and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception.
* Active use of illicit drugs and/or alcohol dependence.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Number (%) of subjects with treatment emergent adverse events (TEAEs) over the study. | 18 months
  Number (%) of subjects with treatment emergent adverse events (TEAEs) over the study, number of TEAEs over the study and rate of TEAEs per subject per Vaso-Occlusive Crisis (VOC) will be summarized overall, by system organ class and by preferred term.
Number (%) of subjects with adjudicated Acute Chest Syndrome (ACS) over the study. | 18 months
  Number (%) of subjects with adjudicated Acute Chest Syndrome (ACS) over the study, number of events of adjudicated ACS and the rates of these events per subject per Vaso-Occlusive Crisis (VOC) will be summarized.
Number (%) of subjects with adjudicated severe and/or generalized cutaneous manifestations over the study | 18 months
  Number (%) of subjects with adjudicated severe and/or generalized cutaneous manifestations over the study, number of events of adjudicated severe and/or generalized cutaneous manifestations and the rates of these events per subject per Vaso-Occlusive Crisis (VOC) will be summarized.
Number (%) of subjects with serious adverse events (SAEs) over the study. | 18 months
  Number (%) of subjects with serious adverse events (SAEs) over the study, number of SAEs over the study and rate of SAEs per subject per VOC will be summarized overall, by system organ class and by preferred term.

SECONDARY OUTCOMES:
Subject re hospitalization | 18 months
  Number (%) of subjects re hospitalized for VOC within 7, 14, and 30 days of most recent discharge will be provided overall. Number of re hospitalizations for VOC within 7, 14, and 30 days of most recent discharge and the rate of re hospitalization for VOC within 7, 14, and 30 days of most recent discharge per subject per VOC will be provided as well.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (96):
- United States (84):
  - University of South Alabama Women's and Children's Hospital, Mobile, Alabama
  - Arkansas Children's Hospital Research Pharmacy, Little Rock, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - UC Davis Medical Center Main Hospital, Sacramento, California
  - University of California Davis Medical Center, Sacramento, California
  - Howard University Center for Sickle Cell disease, Washington D.C., District of Columbia
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Howard University Hospital, Washington D.C., District of Columbia
  - Golisano Childrens Hospital of Southwest Florida, Fort Myers, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - University of Miami, Miami, Florida
  - St. Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta Aflac Cancer and Blood Disorders Center:, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia
  - Emory Children's Center, Atlanta, Georgia
  - Children's Healthcare of Atlanta Aflac Cancer and Blood Disorders Center/, Atlanta, Georgia
  - Children's Healthcare of Atlanta: Scottish Rite Campus, Atlanta, Georgia
  - Memorial Family Medicine Center, Savannah, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - The University of Chicago/Comer Children's Hospital, Chicago, Illinois
  - University of Chicago, Investigational Drug Service Pharmacy, Chicago, Illinois
  - University of Maryland Medical System Investigational Pharmacy, Baltimore, Maryland
  - University of Maryland Medical System, Baltimore, Maryland
  - Johns Hopkins Department of Medicine Clinical Trials Unit, Baltimore, Maryland
  - The Johns Hopkins University School of Medicine, Baltimore, Maryland
  - The Johns Hopkins Hospital Department of Pharmacy Services, Baltimore, Maryland
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Center for Clinical Investigation, Brigham and Women's Hospital, Boston, Massachusetts
  - Investigational Drug Services, Boston, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - University of Mississippi Medical Center - Outpatient Clinical Research Unit, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Center for Outpatient Health, St Louis, Missouri
  - Barnes-Jewish Hospital Department of Pharmacy, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Center for Advanced Medicine, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Bristol Myers Squibb Children's Hospital at Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Kings County Hospital Center, Brooklyn, New York
  - State University of New York (SUNY) Downstate Medical Center, Brooklyn, New York
  - SUNY Downstate Medical Center University Hospital of Brooklyn, Brooklyn, New York
  - Columbia University Medical Center Research Pharmacy, New York, New York
  - MS CHONY Pediatric Emergency Department, New York, New York
  - MS CHONY Pediatric Hematology/Oncology Unit, New York, New York
  - Jacobi Medical Center, The Bronx, New York
  - Duke University Hospital, Investigational Drug Service, Durham, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University Brody School of Medicine, Greenville, North Carolina
  - East Carolina University, Brody School of Medicine, Greenville, North Carolina
  - Leo W. Jenkins Cancer Center, Greenville, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - University of Cincinnati - Hoxworth Building, Cincinnati, Ohio
  - University of Cincinnati Medical Center / Investigational Pharmacy, Cincinnati, Ohio
  - University of Cincinnati Medical Center / Research Office, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University of Cincinnati Physicians Company LLC, Cincinnati, Ohio
  - UC Health Ridgeway Hospital, Cincinnati, Ohio
  - The Ohio State University Investigational Drug Services, Columbus, Ohio
  - The Ohio State University Wexner Center East, Columbus, Ohio
  - The Ohio State University James Comprehensive Cancer Hospital & Solove Research Institute, Columbus, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Hasbro Children's Hospital, Providence, Rhode Island
  - Rhode Island Hospital-Pharmacy Service, Providence, Rhode Island
  - Rhode Island Hospital, Providence, Rhode Island
  - The Miriam Hospital, Providence, Rhode Island
  - Medical University of South Carolina Lifespan Comprehensive Sickle Cell Center, Charleston, South Carolina
  - Medical University of South Carolina-Hospital, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - MUSC Investigational Drug Services, Charleston, South Carolina
  - Cook Children's Hematology and Oncology Center, Fort Worth, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Cook Children's Hematology and Oncology Center-Grapevine, Grapevine, Texas
  - University of Texas Medical School, Houston, Texas
  - Primary Children's Hospital Laboratory, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - Main Hospital-VCU, Richmond, Virginia
  - Virginia Commonwealth University - Investigational Drug Services, Richmond, Virginia
  - Virginia Commonwealth University- Clinical Research Services Unit, Richmond, Virginia
- Canada (12):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Miseracordia Community Hospital, Edmonton, Alberta
  - Kaye Edmonton Clinic 3C, Edmonton, Alberta
  - University of Alberta Hospital, Pharmacy Services, Edmonton, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Research transition Facility, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - The Montreal Children's Hospital / McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dampier CD, Telen MJ, Wun T, Brown RC, Desai P, El Rassi F, Fuh B, Kanter J, Pastore Y, Rothman J, Taylor JG, Readett D, Sivamurthy KM, Tammara B, Tseng LJ, Lozier JN, Thackray H, Magnani JL, Hassell KL; RESET Investigators. A randomized clinical trial of the efficacy and safety of rivipansel for sickle cell vaso-occlusive crisis. Blood. 2023 Jan 12;141(2):168-179. doi: 10.1182/blood.2022015797. PMID 35981565